CLINICAL TRIAL: NCT06494137
Title: Effect of Pre-dosing With Methylcellulose or Psyllium on Colonic Fermentation of Inulin (COCOA3)
Brief Title: Effect of Pre-dosing With Methylcellulose or Psyllium on Colonic Fermentation of Inulin
Acronym: COCOA3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Quadram Institute Bioscience (Other)
Responsible Party: Principal Investigator, Robin Spiller, Professor of Gastroenterology, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FMHS 158-0324
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: inulin; fermentation; colon
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Inulin

STUDY DESIGN:
Intervention Model Description: randomised placebo controlled crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: gels given in opaque plastic bag
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psyllium (Active Comparator): 15g psyllium + 15 inulin dissolved in 250 ml water
  Interventions: Other: inulin
- Methylcelulose (Active Comparator): 15g methylcellulose +15 g inulin dissolved in 250 ml water
  Interventions: Other: inulin
- Maltodextrin (Placebo Comparator): 15g maltodextrin +15 g inulin dissolved in 250 ml water
  Interventions: Other: inulin

INTERVENTIONS:
Other: inulin — inulin from chicory root

SUMMARY:
The aim for this pilot study is to test the hypothesis that pre-dosing with gel-forming dietary fibres (methylcellulose or psyllium) will alter the colonic fermentation of a model fermentable dietary fibre (Inulin) when delivered separately, in contrast to our previous trials where gel-forming and fermentable dietary fibres were co-administered. Performance of each gel-forming dietary fibre will be compared to placebo (water) to assess treatment effectiveness.

DETAILED DESCRIPTION:
4. BACKGROUND AND RATIONALE

The challenge is to understand how various dietary fibres interact to alter colonic fermentation of FODMAPs (fermentable oligosaccharides, disaccharides, monosaccharides and polyols) with the aim of reducing gaseous distension of the colon and hence symptoms. Previous studies 1 have shown how psyllium, a gel forming natural fibre can reduce gas production induced by a dietary FODMAP inulin when it reaches the colon. The investigation will exploiting a range of food grade modified celluloses which can form gels at body temperature to perform human studies to explore whether the beneficial effect of psyllium is unique or will be found with all gelling substances 2.

The mode of action of methylcellulose and psyllium on the reduction in gas production from inulin remains unclear. Possible mechanisms include 1) slowing delivery to the colon by their effect in the small bowel, 2) delayed release of inulin from the dietary fibre gel matrix (i.e. a physical effect) in the colon 3) or a direct effect on the colonic bacteria reducing their production of gas (i.e. a microbiological effect).

References

Aim This pilot study will test the hypothesis that pre-dosing with gel-forming dietary fibres (methylcellulose or psyllium) will alter the colonic fermentation of a model fermentable dietary fibre (Inulin) when delivered separately, in contrast to our previous trials where gel-forming and fermentable dietary fibres were co-administered. Performance of each gel-forming dietary fibre will be compared to placebo (water) to assess treatment effectiveness.

Objective The primary objective of this pilot is to compare the effect of pre-feeding a gel-forming dietary fibre (methylcellulose or psyllium) compared to placebo (water) on the colonic fermentability of Inulin over the six hours immediately post inulin ingestion as assessed from breath hydrogen production.

Secondary Objectives

1. Area under curve (AUC) of breath hydrogen and methane for period 0 - 24hr.
2. Orocecal transit time (OCTT) from breath analysis.
3. Whole gut transit time assessed by blue muffin test.
4. Gas production with in vitro model of colon using participants stool samples (Quadram Institute).
5. Metabolite production (short chain fatty acids) using same in vitro model of colon (Quadram Institute).
6. Analysis of microbiota in participants stool using 16sRNA gene (in collaboration with Quadram Institute).
7. Assessment of habitual dietary FODMAP intake on breath hydrogen response to Inulin

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years old.
* Able to give informed consent.
* Scoring ≤5 (i.e., mild, or less) for symptoms of flatulence, bloating, abdominal pain, loose stool, and hard stool in previous 2 weeks using a modified Gastrointestinal Symptom Rating Scale (5).
* Agrees to consume the meals provided.
* Agrees to not smoke during the breath hydrogen sampling period.

Exclusion Criteria:

* • Pregnancy, lactating, or planning pregnancy during the course of the investigation declared by candidate.

  * History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function.
  * Reported history of previous resection of the oesophagus, stomach, or intestine (excluding appendix).
  * Intestinal stoma.
  * Any medical condition making participation potentially compromising participation in the study e.g., diabetes mellitus, respiratory disease limiting ability to use breath hydrogen analyser, known intolerance to one of the test substances.
  * Has a body mass index (BMI) value less than 18.5 or greater than 35.
  * Will not agree to follow dietary and lifestyle restrictions required.
  * Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors, low dose tricyclic antidepressants, antihistamines, and oral contraceptive pill will be recorded in the CRF but will not be an exclusion criteria).
  * Participants who are taking antibiotics or probiotics as it might alters gut microbiota.
  * Poor understanding of English language.
  * Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM.
  * Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g., cognitive dysfunction, chaotic lifestyle related to substance abuse.
  * Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Breath hydrogen AUC | 0-6 hours
  Area under curve (AUC) from time 0-6 hours (AUC 0-6) of breath hydrogen (ppm.hour) after consumption of inulin intake.

SECONDARY OUTCOMES:
Breath hydrogen AUC | 0-24h
  Area under curve (AUC) from time 0-24hours (AUC 0-24) of breath hydrogen (ppm.hour) after consumption of inulin intake.
Whole gut transit | 0-7days
  Time for blue colour to appear after ingesting muffin labelled with blue food colouring

CONTACTS AND LOCATIONS:
Overall Officials: Robin C Spiller, MD, Principal Investigator — Professor
Locations (1):
- Nottingham Digestive Disease Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gunn D, Abbas Z, Harris HC, Major G, Hoad C, Gowland P, Marciani L, Gill SK, Warren FJ, Rossi M, Remes-Troche JM, Whelan K, Spiller RC. Psyllium reduces inulin-induced colonic gas production in IBS: MRI and in vitro fermentation studies. Gut. 2022 May;71(5):919-927. doi: 10.1136/gutjnl-2021-324784. Epub 2021 Aug 5. PMID 34353864